CLINICAL TRIAL: NCT06933641
Title: Comparison of Paravertebral, Thoracolumbar Interfascial Plane, and Retrolaminar Blocks for Postoperative Analgesia in Lumbar Disc Herniation Surgery: A Randomized Controlled Trial
Brief Title: Regional Blocks for Lumbar Disc Surgery Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Hakan Gokalp TAS, Assistant Professor, Erzincan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-07/06
Record Dates: First submitted 2025-03-26; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Analgesia
Keywords: Lumbar Vertebrae; Postoperative Pain; Nerve Block; Interfascial Plane Blocks; Analgesics, Opioid
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group (No Intervention): All patients received routine intravenous analgesia with 1 g paracetamol and 1 mg/kg tramadol hydrochloride every 12 hours during postoperative ward follow-ups.
- Paravertebral Block Group (Active Comparator): All patients received regional analgesia and routine intravenous analgesia with 1 g paracetamol and 1 mg/kg tramadol hydrochloride every 12 hours during postoperative ward follow-ups.
  Interventions: Procedure: Regional Analgesia
- Thoracolumbar Interfascial Plane Block Group (Experimental): All patients received regional analgesia and routine intravenous analgesia with 1 g paracetamol and 1 mg/kg tramadol hydrochloride every 12 hours during postoperative ward follow-ups.
  Interventions: Procedure: Regional Analgesia
- Retrolaminar Block Group (Experimental): All patients received regional analgesia and routine intravenous analgesia with 1 g paracetamol and 1 mg/kg tramadol hydrochloride every 12 hours during postoperative ward follow-ups.
  Interventions: Procedure: Regional Analgesia

INTERVENTIONS:
Procedure: Regional Analgesia — 20 cc of local anesthetic solution, comprising 10 cc of 0.5% bupivacaine and 10 cc of 0.9% NaCl bilaterally, was injected into each side once
  Arms: Paravertebral Block Group; Retrolaminar Block Group; Thoracolumbar Interfascial Plane Block Group

SUMMARY:
Objective The goal of this prospective randomized controlled experiment was comparing the analgesic efficacy, opioid needs, and adverse effect profiles of Paravertebral Block (PVB), Thoracolumbar Interfascial Plane Block (TLIP), and Retrolaminar Block (RLB) in patients undergoing lumbar disc herniation surgery.

Methods 180 adults (ASA I-III) undergoing elective lumbar disc herniation surgery made up this single-center study. Among the exclusion criteria were coagulation problems, injection site infection, allergy to local anesthetics, and incapacity to provide informed consent. Patients were randomly assigned into four groups: Control (systemic analgesia only), PVB, TLIP, and RLB (45 patients per group). An expert anesthesiologist supervised the ultrasonography during each block. The Visual Analog Scale (VAS) was used to measure postoperative pain at 0, 1, 2, 6, 12, and 24 hours after surgery. This was the primary outcome. Motor block incidence, rescue morphine consumption, and Quality of Recovery-40 (QoR-40) scores at 24 hours were secondary objectives. Unfavorable incidents were noted. ANOVA and Kruskal-Wallis tests (p<0.05) were used to examine the data.

DETAILED DESCRIPTION:
With an annual frequency of 10% to 15% among healthy adults, low back pain is a significant global public health concern. For low back pain, the typical visual analog scale (VAS) score is approximately 4, indicating moderate pain severity (1). A common cause of back and leg pain is intervertebral disc herniation, which causes throbbing anguish in the lower extremities along with radicular pain. Lumbar disc surgery is a common procedure for people with moderate to severe back pain and radicular symptoms. Surgery may be necessary for people with chronic symptoms, neurological deficits, or inadequate pain relief with conservative treatment, even though acute intervertebral disc herniation often resolves on its own without surgery.

After lumbar disc herniation surgery, postoperative pain management is still crucial since inadequate pain management can lead to prolonged hospital stays, slower recovery, and a poorer quality of life. Numerous strategies have been used to manage postoperative pain, such as regional anesthetic procedures, epidural steroid injections, nonsteroidal anti-inflammatory drugs (NSAIDs), and even unconventional methods like electroacupuncture. Due of their capacity to provide targeted pain relief while minimizing systemic effects, regional anesthetic procedures have become increasingly popular among these.

In lumbar surgery, the paravertebral block (PVB) is a common regional anesthetic technique. A local anesthetic is injected close to the spinal nerves, and it typically relieves pain over four dermatomes (two above and two below the injection site). Patients with spinal anomalies or those for whom neuraxial anesthesia is contraindicated have been shown to benefit greatly from PVB. Additionally, it differs from other peripheral nerve blocks in its ability to reduce visceral and somatic pain. However, PVB requires technical know-how and might have negative effects like vascular injury and pneumothorax, particularly when performed by unskilled professionals.

PVB is being replaced by more recent truncal block methods such retrolaminar blocks (RLB) and the thoracolumbar interfascial plane (TLIP). For effective analgesia during lumbar spine surgery, the TLIP block targets the thoracolumbar fascia. According to recent studies, the TLIP block can enhance recovery quality, decrease postoperative pain levels, and lessen the need for rescue medications. In a similar vein, the RLB, which involves administering a local anesthetic into the retrolaminar area, has been associated with shorter recovery periods, reduced postoperative pain scores, and decreased narcotic usage. Compared to PVB, these contemporary techniques are less invasive, simpler to do under ultrasound guidance, and possibly less problematic.

Comparative research is required to evaluate the effectiveness, safety, and viability of TLIP and RLB in the setting of lumbar disc herniation surgery, given their increasing popularity as PVB substitutes. Previous research has primarily focused on the individual efficacy of these methods; however, head-to-head comparisons remain limited. The aim of this study is to investigate at the analgesic efficacy, sensory coverage, and side effect profiles of PVB, TLIP, and RLB in patients having lumbar disc herniation surgery. By doing so, we intend to determine if TLIP and RLB are viable alternatives to PVB, particularly in terms of side effects and patient recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 65 who were having elective lumbar disc herniation surgery and had ASA I-III ratings made up the study

Exclusion Criteria:

* The study excluded patients having a history of opioid dependency, coagulation issues, difficult behavior, pharmaceutical allergies, prior spinal surgery, or unwillingness to participate in the experiment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 0 hour, 1 hour, 2 hour, 6 hour, 12 hour, 24 hour after surgery
  The pain is scaled with Visual Analogue Scale score in 4 groups

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gökalp Taş, Study Director — Erzincan Binali Yildirim Universitesi
Locations (1):
- Erzincan University, Erzincan, Merkez, Turkey (Türkiye)